CLINICAL TRIAL: NCT05249426
Title: An Open Label Trial of BI 765063 in Combination With BI 754091 (Ezabenlimab) Alone or With BI 836880, Chemotherapy, or Cetuximab, in Patients With Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma (HNSCC) or Hepatocellular Carcinoma (HCC)
Brief Title: A Study to Test Whether Different Combinations of BI 765063, Ezabenlimab, Chemotherapy, Cetuximab, and BI 836880 Help People With Head and Neck Cancer or Liver Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1443-0002; 2021-003473-59 (EudraCT Number)
Record Dates: First submitted 2022-02-10; First posted 2022-02-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Squamous Cell Carcinoma (HNSCC)
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab

STUDY DESIGN:
Masking Description: Partly randomized trial. Patients will be randomized into cohort A, B, C and D. No randomization in cohort E.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort A: BI 765063 + ezabenlimab + cetuximab (Experimental): 30 Signal Regulatory Protein Alpha (SIRPα) V1/V1 homozygous patients with 2nd line recurrent/metastatic Head and Neck Squamous Cell Carcinoma (HNSCC) who had received prior platinum-based therapy within the recurrent/metastatic setting.
  Interventions: Drug: BI 765063; Drug: Ezabenlimab; Drug: Cetuximab
- Cohort B: BI 765063 + ezabenlimab + chemo (invest choice) (Experimental): 30 SIRPα V1/V1 homozygous patients with 2nd line recurrent/metastatic HNSCC who had received prior platinum-based therapy within the recurrent/metastatic setting.
  Interventions: Drug: BI 765063; Drug: Ezabenlimab; Other: Investigator´s Choice Chemotherapy
- Cohort C: BI 765063 + ezabenlimab (Experimental): 30 SIRPα V1/V1 homozygous patients with advanced or metastatic 1st line Hepatocellular Carcinoma (HCC).
  Interventions: Drug: BI 765063; Drug: Ezabenlimab
- Cohort D: BI 765063 + ezabenlimab + BI 836880 (Experimental): 30 SIRPα V1/V1 homozygous patients with advanced or metastatic 1st line HCC.
  Interventions: Drug: BI 765063; Drug: Ezabenlimab; Drug: BI 836880
- Cohort E: BI 765063 + ezabenlimab + BI 836880 (Experimental): 30 SIRPα V1/V1 homozygous patients with advanced or metastatic 2nd line HCC who progressed on therapy with atezolizumab in combination with bevacizumab.
  Interventions: Drug: BI 765063; Drug: Ezabenlimab; Drug: BI 836880

INTERVENTIONS:
Drug: BI 765063 — BI 765063 (anti-Signal Regulatory Protein Alpha (SIRPα) Monoclonal Antibody (mAb))
Drug: Ezabenlimab — Ezabenlimab (anti-Programmed cell death protein 1 (PD-1) Monoclonal Antibody (mAb))
  Other Names: BI 754091
Drug: BI 836880 — BI 836880 (anti-Vascular Endothelial Growth Factor (VEGF) / Angiopoetin 2 (Ang2))
  Arms: Cohort D: BI 765063 + ezabenlimab + BI 836880; Cohort E: BI 765063 + ezabenlimab + BI 836880
Drug: Cetuximab — Cetuximab
  Arms: Cohort A: BI 765063 + ezabenlimab + cetuximab
Other: Investigator´s Choice Chemotherapy — Allowable chemotherapies include: paclitaxel, docetaxel, capecitabine, 5-fluorouracil, methotrexate or combinations thereof
  Arms: Cohort B: BI 765063 + ezabenlimab + chemo (invest choice)

SUMMARY:
With an amendment of the protocol, this study is only open to adults with head and neck cancer. Previously also adults with liver cancer joined. This is a study for people for whom previous treatment was not successful or no standard treatment exists. The purpose of this study is to find out whether combining different medicines make tumours shrink.

The tested medicines in this study are antibodies that act in different ways against cancer. BI 765063 and ezabenlimab may help the immune system fight cancer (checkpoint inhibitors). Cetuximab blocks growth signals and may prevent the tumour from growing. BI 836880 blocks the formation of new blood vessels that the tumour needs to grow.

With amendments of the protocol, all participants receive cetuximab in addition to BI 765063 and ezabenlimab. Ezabenlimab treatment and any other assigned treatment are given no longer than 2 years. Previously, BI 765063 and ezabenlimab were also given alone, or in combination with chemotherapy, or with BI 836880. BI 765063, ezabenlimab, and BI 836880 are given as infusions into veins every 3 weeks. Cetuximab is given as an infusion every 1 or 2 weeks. Participants can stay in the study as long as they benefit from treatment and can tolerate it. They regularly visit the study site where doctors check participants' health and take note of any unwanted effects. The doctors also monitor the size of the tumour.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF) prior to any trial-specific procedures.
* Male or female aged ≥ 18 years at the time of ICF signature.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at the screening visit.
* Expected life expectancy of at least 3 months.
* Patients homozygous for V1 allele (including V1-like alleles) of Singal Regulatory Protein-alpha (SIRPα) (V1/V1 SIRPα genotype). SIRPα polymorphism will be assessed in blood sampling (using patient Deoxyribonucleic Acid [DNA]) during Screening 1 Visit.
* Patients with at least one measurable lesion as per Response Evaluation Critiera In Solid Tumours (RECIST) version 1.1 (v1.1).
* Patients must agree to provide a mandatory pre-treatment (baseline) biopsy and an ontreatment fresh tumour biopsy (unless medically contraindicated. or mandatory requirement is lifted by the sponsor). Details on biopsy sample collection are provided in the Lab Manual.

  -- Pre-treatment (baseline) biopsy: A fresh tumour biopsy before receiving the trial medication is preferred. In case a fresh tumour biopsy cannot be obtained, the Sponsor must be notified and archival formalin-fixed paraffin embedded (FFPE) tumour tissue block from the most recent time point before entering the trial must be provided (maximum 6 months prior to study entry). If these requirements cannot be met, the patient may still be allowed to enter the study at the discretion of the sponsor, after discussion between the Investigator and Sponsor.
* Female patients. Women of childbearing potential (WOCBP) must agree to use highly effective methods of contraception per ICH M3 (R2), that results in a less than 1% per year failure rate when used consistently and correctly, starting at the screening visit, during the trial and for 6 months after the end of trial treatment. The requirement of contraception does not apply to women of no childbearing potential, but they must have evidence of such at screening. Women of childbearing potential must have a serum negative pregnancy test within 72 hours prior to first drug administration.

Women who are postmenopausal for at least 1 year (defined as more than 12 months since last menses) or are surgically sterilized do not require this test. The following methods of contraception are considered highly effective:

* Combined (oestrogen and progestogen containing) hormonal birth control that prevents ovulation (oral, intravaginal, transdermal)
* Progestogen-only hormonal birth control that prevents ovulation (oral, injectable, implantable)
* Intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
* Bilateral tubal occlusion
* Vasectomised partner (provided that this is the sole sexual partner and has received medical assessment of the surgical success)
* Sexual abstinence (if accepted by local ethics boards and regulatory agencies as highly effective) Sexual abstinence is defined as refraining from heterosexual intercourse during the entire study period from screening through 6 months after last trial treatment. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject.

Periodic abstinence (calendar, symptothermal, post-ovulation methods) is not an acceptable method of contraception for use during this trial.

Although use of a contraceptive pill and Intrauterine device (IUD) together are considered a highly- effective method of birth control, women of childbearing potential taking a contraceptive pill must use an additional barrier method for the entire duration of the trial treatment intake and for 6 months after the end of the trial treatment intake. WOCBP is defined as: fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. Tubal ligation is NOT a method of permanent sterilisation. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.

Further inclusion criteria apply.

Exclusion criteria:

* Patients with at least one SIRPα V2 allele, i.e. SIRPα V1/V2 or V2/V2 individuals.
* Patients with symptomatic/active central nervous system (CNS) metastases. Patients with previously treated brain metastases are eligible, if there is no evidence of progression for at least 28 days before the first trial drug administration without requirement for treatment with corticosteroids, as ascertained by clinical examination and brain imaging (MRI (magnetic resonance imaging) or CT (computed tomography)) during the screening period.
* Prior allogeneic stem cell or solid organ transplantation.
* Any tumour location necessitating an urgent therapeutic intervention (e.g., palliative care, surgery or radiation therapy, such as spinal cord compression, other compressive mass, uncontrolled painful lesion, bone fracture).
* Presence of active invasive cancers other than the one treated in this trial within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin, or in situ carcinoma of uterine cervix, or other local tumours considered cured by local treatment.
* Patients with active autoimmune disease or a documented history of autoimmune disease, that requires systemic treatment, i.e. corticosteroids or immunosuppressive drugs, except patients with vitiligo, resolved childhood asthma/atopy, alopecia, or any chronic skin condition that does not require systemic therapy; patients with autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone and/or controlled Type 1 diabetes mellitus on a stable insulin regimen are eligible.
* History of severe hemorrhagic or thromboembolic event in the past 12 months (excluding central venous catheter thrombosis, peripheral deep vein thrombosis and portal vein thrombosis due to HCC tumor invasion).
* Known prior history of severe infusion related reactions to monoclonal antibodies (Grade ≥ 3 National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events (CTCAE) v5.0).

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response (OR) | Up to 24 months.
  Objective response (OR) with confirmation, defined as the best overall response of complete response (CR) or partial response (PR), where best overall response is determined according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1 (v1.1) by investigator's assessment from first treatment administration until the earliest of disease progression, death, or last evaluable tumour assessment before start of subsequent anti-cancer therapy, lost to follow-up or withdrawal of consent.

SECONDARY OUTCOMES:
Occurrence of treatment emergent adverse events (AEs) | Up to 24 months.
  Occurrence of treatment emergent adverse events (AEs) by investigator's assessment from first treatment administration until the earliest of death, subsequent anti-cancer therapy, lost to follow-up or withdrawal of consent.
Duration of objective response (DOR) | Up to 24 months.
  Duration of objective response (DOR), defined as the time from first documented complete response (CR) or partial response (PR) (RECIST v1.1) until the earliest of progressive disease (PD) or death among patients with objective response (OR).
Disease control (DC) | Up to 24 months.
  Disease control (DC), defined as best overall response of complete reponse (CR), partial reponse (PR), or stable disease (SD) where best overall response is defined according to RECIST v1.1 as assessed by the Investigator until the earliest of disease progression, death, or last evaluable tumour assessment before start of subsequent anti-cancer therapy, or permanent treatment discontinuation.
Progression-free survivial (PFS) | Up to 24 months.
  Progression-free survival (PFS), defined as the time from first treatment administration until progressive disease (PD) according to RECIST v1.1 or death from any cause, whichever occurs earlier.

CONTACTS AND LOCATIONS:
Locations (25):
- Valkyrie Clinical Trials, Los Angeles, California, United States
- France (6):
  - CTR Georges-François Leclerc, Dijon
  - CTR Leon Berard, Lyon
  - HOP Timone, Marseille
  - INS Curie, Paris
  - HOP Civil, Strasbourg
  - INS Claudius Regaud IUCT-Oncopole, Toulouse
- Japanese Foundation for Cancer Research, Tokyo, Koto-ku, Japan
- Malaysia (2):
  - Hospital Sultan Ismail, Johor Bahru
  - Sarawak General Hospital, Kuching, Sarawak
- Mexico (3):
  - ARKE SMO S.A. de C.V, Mexico City
  - FAICIC S de RL de C.V., Veracruz
  - Investigacion Biomedica para el Desarrollo de Farmacos, S.A. de C.V., Zapopan
- ARENSIA Exploratory Medicine, Chisinau, Moldova
- Mandziuk Slawomir Specialist Medical Practice, Lublin, Poland
- Romania (2):
  - "Prof. Dr. Alexandru Trestioreanu" Oncology Institut, Bucharest
  - Institutul Oncologic "Prof. Dr. Ion Chiricuta", Cluj-Napoca
- Spain (3):
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital Clínico San Carlos, Madrid
- Thailand (2):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Songklanagarind Hospital, Songkhla
- United Kingdom (3):
  - King's College Hospital, London
  - The Royal Marsden Hospital, Chelsea, London
  - Hammersmith Hospital, London

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com